CLINICAL TRIAL: NCT04453176
Title: Evaluation of the Satisfaction of Patients Coming "on Foot" in the Operating Room (Standing, Dignified, Relaxed)
Brief Title: Evaluation of the Satisfaction of Patients Coming "on Foot" in the Operating Room
Acronym: Bloc3D
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2018/PC-01
Record Dates: First submitted 2020-01-27; First posted 2020-07-01 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Anesthesiology; Satisfaction, Patient; Surgery
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- operating block admission "on foot": Patient going to the oparating block on foot
  Interventions: Other: Patient Satisfaction
- standard operating block admission: Patient going to the operating room in a conventional way (stretcher)
  Interventions: Other: Patient Satisfaction

INTERVENTIONS:
Other: Patient Satisfaction — Patient satisfaction evaluated with EVAN G questionnaire

SUMMARY:
Ambulatory surgery is currently experiencing unprecedented growth and is becoming the standard of care compared to traditional hospitalization. Without mentioning the obvious financial gains, the benefits of ambulatory care essentially lie in optimised perioperative comfort. This comfort is due to a limited period of stay (< 12 hours) and to the proactive action of the care providers.

In this context, the optimization of the whole patient's journey during the perioperative period has been reviewed and adapted to personalized management within healthcare facilities. For more than a year now, multimodal approaches such as early rehabilitation have been undertaken, including

* morning admission with an innovative principle of "3D" patient (standing, dignified, relaxed)
* no premedication, wearing glasses and wigs,
* Drinking on the morning of the intervention (2H before admission),
* Walking to the block on foot (or in a wheelchair), return adapted to the wheelchair and no longer in a stretcher,
* fast resumption of feeding.

Currently, in the investigator's various institutions, several modes of transport to the operating theatres coexist. The purpose of this observational study is to evaluate this optimization of perioperative management "3D mode", in particular the mode of transport.

The main objective is to determine the level of patient satisfaction with this management using a standardized quality questionnaire: the "EVAN" questionnaire. This questionnaire contains 22 items allowing a global analysis of patient satisfaction. This questionnaire is already routinely conducted in many institutions. The EVAN questionnaire will be supplemented by questionnaires assessing the level of perioperative anxiety. They will be initiated into the anesthesia consultation, and finalized on the day of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yars
* Consent to participate

Exclusion Criteria:

* Emergency surgery
* ASA >4
* Difficulties in French reading, incapacity to complete questionnaire
* patient in a wheelchair or stretcher or having difficulty walking alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study are patients at least 18 years old, hospitalized for scheduled surgery, who have accepted the principle of the study, are able to complete the EVAN-G questionnaire and are able to walk alone.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Satisfaction of day case surgery: EVAN-G score | Day 0
  Satisfaction is measured with an EVAN-G score (1-100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Fayard, MD, Principal Investigator — CHU Nimes, France
Locations (5):
- France (5):
  - CHU Nimes, Nîmes, Gard
  - Clinique Juge, Marseille
  - Institut paoli Calmette, Marseille
  - Chu Montpellier - Saint-Eloi, Montpellier
  - Institut de cancerologie de Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No